CLINICAL TRIAL: NCT02693652
Title: A Single Center, Open Labeled Phase I/IIa Study to Evaluate Safety, Tolerability and Efficacy of a Therapeutic Hepatitis B Vaccine in Oral Antiviral Drug-treated Chronic Hepatitis B Virus Carriers
Brief Title: A Study to Evaluate the Safety and Efficacy of Therapeutic Hepatitis B Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CHA Vaccine Institute Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVI-HBV-002-CT1301
Record Dates: First submitted 2016-02-18; First posted 2016-02-29 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CVI-HBV-002 (20ug, 3 shots) (Experimental): * HBV surface antigen 20ug/dose
  * Intramuscular injection at 0, 1, 2 month
  Interventions: Biological: CVI-HBV-002
- CVI-HBV-002 (20ug, 6 shots) (Experimental): * HBV surface antigen 20ug/dose
  * Intramuscular injection at 0, 1, 2, 3, 4, 5 month
  Interventions: Biological: CVI-HBV-002
- CVI-HBV-002 (40ug, 3 shots) (Experimental): * HBV surface antigen 40ug/dose
  * Intramuscular injection at 0, 1, 2 month
  Interventions: Biological: CVI-HBV-002
- CVI-HBV-002 (40ug, 6 shots) (Experimental): * HBV surface antigen 40ug/dose
  * Intramuscular injection at 0, 1, 2, 3, 4, 5 month
  Interventions: Biological: CVI-HBV-002

INTERVENTIONS:
Biological: CVI-HBV-002 — * Investigational product: CVI-HBV-002
  * Dose: 20ug or 40ug
  * Frequency: 3 or 6 times
  * Vaccination schedule: 0, 1, 2 months or 0, 1, 2, 3, 4, 5 months
  * Administration route: Intramuscular injection

SUMMARY:
A single center, open labeled phase I/IIa study to evaluate safety, tolerability and efficacy of a therapeutic hepatitis B vaccine in oral antiviral drug-treated chronic hepatitis B virus carriers

DETAILED DESCRIPTION:
* Objectives: To explore the appropriate dose of a therapeutic hepatitis B vaccine through the evaluation of safety, tolerability, and efficacy
* Subjects: Chronic hepatitis B carrier with normal ALT range
* Study hypothesis: The immune tolerance break and strong immune responses in the chronic hepatitis B carrier could be achieved with therapeutic hepatitis B vaccine containing novel adjuvant

ELIGIBILITY:
Inclusion Criteria:

1. Adult between 19 to 60 years of age
2. Chronic hepatitis B carriers (HBsAg positive over 6 months)
3. HBeAg positive patient, or patient who had lost HBeAg during Antiviral drug treatment
4. Antiviral drug treated patient reducing the HBV DNA level below 2000 IU/mL measured by COBAS TaqManM HBV Test (Duration of drug administration should be over 6 months and no limitation on the type of antiviral drug)
5. Patient has low ALT than 1.1 fold of upper limit of normal ALT level at screening
6. Patient is able to provide written informed consent by oneself or legal representative

Exclusion Criteria:

1. Patient has liver diseases except chronic hepatitis B (i.e. hematochromatosis, alcoholic liver disease, nonalcoholic fatty liver disease, alpha-1 antitrypsin deficiency etc.)
2. Patient has one or more test results and symptoms at the screening

   * ALT > upper limit of normal level X 1.1
   * Total bilirubin > upper limit of normal
   * Prothrombin time > Over 3 second than normal
   * Serum Albumin < 30 g/L (3 g/dL)
   * Patient has history of ascites, yellow jaundice, variceal hemorrhage, hepatic encephalopathy, or liver failure
   * Liver FibroScan > F3 (F0: no fibrosis, F1: portal fibrosis, F2: periportal fibrosis, F3: septal fibrosis, F4: cirrhosis)
3. Patient has one or more test results at the screening

   * Hemoglobin < 9.0 g/dL
   * Absolute neutrophil count (ANC) < 1.5 x 109 /L (1500 /mm3)
   * Platelet count < 100 x 109 /L (100 x 103 /mm3)
   * Serum creatinine > 1.5 mg/dL
   * Serum amylase > 2 x ULN and Lipase > 2 x ULN
4. Patient has history of Interferon treatment
5. Patient is pregnant or breastfeeding or intending to become pregnant during the study
6. Patient has active microbial, viral, or fungal infections in need of systemic treatment
7. Alpha-fetoprotein (AFP) > 50 ng/mL or Hepatocellular Carcinoma (HCC) patient
8. Among the patients treated with immunosuppressive drug within 6 months before screening, suspected case of the declined immunity in the opinion of the investigator
9. Patient had long term systemic treatment (more than 14 days consecutively) of high dose (over 20 mg of prednisolone or equivalent dose*) corticosteroid (Decision to participate of patient who had local treatment of corticosteroid is allowed in the opinion of the investigator)

   *equivalent to cortisone 125 mg, hydrocortisone 100 mg, prednisone 20 mg, methylprednisolone 16 mg, triamcinolone 16 mg, dexamethasone 3 mg, or betamethasone 2.4 mg
10. Patient diagnosed with a malignant tumor within 5 years before screening or relapsed patient (Benign tumor patient is able to participate in this study at the discretion of the investigator)
11. Patient has history of organ transplantation
12. Patient has serious disease judged by investigator such as heart failure, renal failure, and pancreatitis
13. Patient has history of serious heart disease (NYHA Functional Class III or IV heart failure, myocardial infarction within 6 months, treatment required ventricular tachyarrhythmias, or unstable angina etc.)
14. Patient has seizure disorder required anticonvulsants treatment
15. Uncontrollable diabetic patient (FBS>130mg/dl, HbA1c>7.5%)
16. Uncontrollable hypertension patient (SBP≥140mmHg 또는 DBP≥90mmHg)
17. HCV, HDV, or HIV patient
18. Patient has a plan to participate in other clinical study, or took part in other clinical study within 1 month before enrollment
19. Patient has hypersensitivity or anaphylactic reaction for components of investigational product or HBV vaccine
20. Patient has continuous drinking (>21 units/week, 1 unit = 10g of pure alcohol) or dependence on alcohol
21. Patient concerned about the decline in daily activity or not able to understand the objectives and methods due to the psychiatric problems
22. Patient has potential to severe febrile or systemic reaction
23. Subject unacceptable in this study under the opinion of the investigator

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2017-08-22 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (including incidence of adverse events or expected adverse reactions for vaccine treatment) measured for 7 days after each vaccination | 7 days after each vaccination
  Occurrence of severe local and/or systemic tolerability signs and symptoms measured for 7 days after each vaccination

SECONDARY OUTCOMES:
HBeAg loss | at the 3rd and 5th month (for 3 shot group) or 6th and 8th month (for 6 shot group)
  HBeAg disappearance at the 3rd and 5th month (for 3 shot group) or 6th and 8th month (for 6 shot group) comparing with that of baseline
HBe seroconversion rate | at the 3rd and 5th month (for 3 shot group) or 6th and 8th month (for 6 shot group)
  HBeAg seroconversion rate at the 3rd and 5th month (for 3 shot group) or 6th and 8th month (for 6 shot group) comparing with that of baseline
HBsAg loss | at the 3rd and 5th month (for 3 shot group) or 6th and 8th month (for 6 shot group)
  HBsAg disappearance at the 3rd and 5th month (for 3 shot group) or 6th and 8th month (for 6 shot group) comparing with that of baseline
HBsAg seroconversion rate | at the 3rd and 5th month (for 3 shot group) or 6th and 8th month (for 6 shot group)
  HBsAg seroconversion rate at the 3rd and 5th month (for 3 shot group) or 6th and 8th month (for 6 shot group) comparing with that of baseline
HBV specific T cell immunity | at the 3rd month (for 3 shot group) or 6th month (for 6 shot group)
  HBV specific T cell response at the 3rd month (for 3 shot group) or 6th month (for 6 shot group) comparing with that of baseline
HBV DNA level | at the 3rd and 5th month (for 3 shot group) or 6th and 8th month (for 6 shot group)
  HBV DNA level at the 3rd and 5th month (for 3 shot group) or 6th and 8th month (for 6 shot group) comparing with that of baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Rim, M.D., Ph.D., Principal Investigator — Bundang CHA General Hospital
Locations (1):
- Bundang CHA General Hospital, Seongnam-si, Gyeonggi-do, South Korea